CLINICAL TRIAL: NCT00445016
Title: Neurologic Complications in Peripheral Regional Anesthesia - A Clinical Follow Up Study to Evaluate the Incidence of Neurologic Complications Defined According to a Standardized Protocol Considering Motoric and Sensory Function and Pain
Brief Title: Neurologic Complications in Peripheral Regional Anesthesia - An Evaluation Based on a Standardized Protocol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: BG Unfallklinik Murnau (Other)
Responsible Party: Dr Michael Neuburger, BG Unfallklinik Murnau
Other Study IDs: nd001
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Anesthesia, Conduction; Nerve Block; Adverse Effects
Keywords: peripheral regional anesthesia; nerve damage; adverse effects; neurologic complication; neuropathy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: peripheral regional anesthesia — evaluation and description of adverse effects

SUMMARY:
To evaluate the incidence of neurologic complications as a consequence of peripheral regional anesthesia, all patients receiving peripheral nerve blocks will be evaluated according to a standardized protocol screening pain, motoric and sensory function recovering to defined periods, and according to a study protocol defining the items.

DETAILED DESCRIPTION:
Neurologic complications as an adverse effect occur in all types of regional anesthesia. Reviewing the literature, the incidence spreads from 0.02 up to 3 percent. The incidence remains unclear because of different types of definitions, too. In this study, we evaluate all patients receiving peripheral regional anesthesia 24 hours after block performance according to a standardized study protocol. In case of any conspicuousness concerning motoric or sensory function or pain, the patient will be evaluated again after 48 hours. Further on, in case of neurologic dysfunction, periods of investigation will be after 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months and 1 year. This study includes the definition for nerve damage concerning motoric and sensory neural function and pain.

The patients will be recruited among all patients from our hospital receiving continuous peripheral regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving peripheral regional anesthesia

Exclusion Criteria:

* Missing agreement

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving peripheral regional anesthesia (routine)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-05; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Buettner, MD, Study Chair — BG Unfallklinik Murnau
Locations (1):
- BG Unfallklinik, Murnau am Staffelsee, Bavaria, Germany

REFERENCES:
- See also: Related Info — http://www.bgu-murnau.de